CLINICAL TRIAL: NCT02011529
Title: A Team Approach to Improve the Quality of Diabetes Care for Patients With Schizophrenia
Brief Title: TEAMcare for Diabetes in Mental Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lydia Chwastiak, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44422-G; R21DK096286-01A1 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-13 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEAMcare treatment of diabetes (Active Comparator)
  Interventions: Other: TEAMcare treatment of diabetes
- Treatment as usual (No Intervention): Participants randomized to treatment as usual will receive their usual mental health treatment and primary care treatment

INTERVENTIONS:
Other: TEAMcare treatment of diabetes — TEAMcare is an evidence-based collaborative care approach to the treatment of diabetes and psychiatric illness. It involves structured visits with a study nurse to monitor psychiatric symptoms, control of medical disease, and self-care activities. The nurses use motivational coaching to help patients solve problems and set goals for improved self-care and medication adherence. Medications for diabetes, hypertension, and hyperlipidemia are monitored and therapy intensified based on treat-to-target guidelines. All of these process and outcome measures are tracked in a registry designed for the study, and the nurses receive weekly supervision with a psychiatrist, an endocrinologist and a psychologist in order to review new cases and to track progress. Once a patient achieves targeted levels for relevant measures, the patient and the nurse develop a maintenance plan.
  Arms: TEAMcare treatment of diabetes

SUMMARY:
This proposal aims to demonstrate the feasibility and acceptability of adapting TEAMcare for patients with schizophrenia. The aim of this innovative mental health center-based team intervention is to improve diabetes, cardiovascular and psychiatric outcomes among patients with poorly controlled type 2 diabetes. The study will be conducted in two phases over the 2-year grant period.

Phase 1. Development of the adapted TEAMcare intervention and training of team members.

Phase 2. During year 2, we will implement the intervention on the caseload of 40 outpatients at Harborview Mental Health Services with schizophrenia and poorly controlled type 2 diabetes. The intervention involves the management of subjects' diabetes, hypertension, and hyperlipidemia by a CMHC diabetes team for 6 months (advanced nurse specialist on-site at supervised in weekly meetings by a psychiatrist and a UW Diabetes Center endocrinologist).

The primary aim of this pilot research grant is to evaluate the feasibility of implementing this complex intervention, in order to guide the design of a larger scale efficacy study (R01). Both process and outcome measures will be evaluated at baseline, and at 3- and 6-month follow-up visits for the 40 subjects enrolled in this feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

* adult (18-70 years);
* enrolled to receive mental health treatment at Harborview Mental Health Services or Downtown Emergency Services Mental Health center
* a diagnosis of type 2 diabetes mellitus or cardiovascular disease
* Hemoglobin A1c >8 or BP > 140/90

Exclusion Criteria:

* cognitive, hearing, or language impairment that would preclude a subject from providing informed consent;
* current suicidality, homicidality, or grave disability that requires psychiatric hospitalization;
* current substance abuse or dependence, as defined by SCID.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months

SECONDARY OUTCOMES:
Blood Pressure | 6 months
LDL cholesterol | 6 months

OTHER OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Chwastiak, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Ludman EJ, Young B, Peterson D, Rutter CM, McGregor M, McCulloch D. Collaborative care for patients with depression and chronic illnesses. N Engl J Med. 2010 Dec 30;363(27):2611-20. doi: 10.1056/NEJMoa1003955. PMID 21190455
- [Derived] Chwastiak LA, Luongo M, Russo J, Johnson L, Lowe JM, Hoffman G, McDonell MG, Wisse B. Use of a Mental Health Center Collaborative Care Team to Improve Diabetes Care and Outcomes for Patients With Psychosis. Psychiatr Serv. 2018 Mar 1;69(3):349-352. doi: 10.1176/appi.ps.201700153. Epub 2017 Dec 1. PMID 29191136